CLINICAL TRIAL: NCT03946800
Title: A Phase 1, Open-label, Dose-escalation and Expansion Study of MEDI1191 Administered Intratumorally as Monotherapy and in Combination With Durvalumab in Subjects With Advanced Solid Tumors
Brief Title: A Study of MEDI1191 in Sequential and Concurrent Combination With Durvalumab in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D8510C00001; 2020-005784-31 (EudraCT Number)
Record Dates: First submitted 2019-05-06; First posted 2019-05-13 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Solid Tumors; Cancer
Keywords: MEDI1191; Durvalumab; MEDI4736; Imfinzi
MeSH Terms: conditions — Neoplasms | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MEDI1191 escalation in combination with durvalumab (Experimental): MEDI1191 escalation in sequential and concurrent combination with durvalumab
  Interventions: Biological: MEDI1191; Biological: Durvalumab
- MEDI1191 expansion in combination with durvalumab (Experimental): MEDI1191 expansion in concurrent combination with durvalumab
  Interventions: Biological: MEDI1191; Biological: Durvalumab

INTERVENTIONS:
Biological: MEDI1191 — Subjects will receive MEDI1191 (at least twice)
Biological: Durvalumab — Subject will receive durvalumab every 4 weeks

SUMMARY:
To evaluate MEDI1191 administered intratumorally in sequential and concurrent combination with intravenous durvalumab in patients with solid tumors.

DETAILED DESCRIPTION:
This is a multicenter, open-label study to evaluate MEDI1191 delivered by intratumoral injection in sequential and concurrent combination with intravenous durvalumab to subjects with solid tumors. The study has a dose escalation design using mTPI-2 to evaluate a range of doses.

ELIGIBILITY:
Inclusion Criteria:

* ECOG 0 to 1.
* Adequate organ function within 2 weeks of starting study treatment.
* Prior to the first dose of MEDI1191, subjects with central nervous system (CNS) metastases must have been treated and must be asymptomatic.
* Cessation of systemic corticosteroids at doses exceeding 12 mg/day prednisone or equivalent, methotrexate, azathioprine, ustekinumab (Stelara®), and tumor necrosis factor (TNF)-α/IL-6 blockers for at least 7 days prior to the first dose of MEDI1191.
* Subjects must have at least one lesion suitable for intratumoral dosing for superficial lesions but at least two lesion suitable for intratumoral dosing for deep-seated lesions.
* Subjects must have at least one non-injected lesion that can be measured by RECIST v1.1.
* Histologic or cytologic confirmation of advanced solid tumor.
* Received and have progressed on or refractory to at least 1 line of standard systemic therapy in the recurrent/metastatic setting.
* Highly effective method of contraception from screening, and must agree to continue using such precautions for 3 months after the final dose of investigational product.
* Nonsterilized male subjects who are sexually active with a female partner of childbearing potential must use a male condom with spermicide from Day 1 through 3 months after receipt of the final dose of investigational product.

Exclusion Criteria:

* Subjects who have received prior IL-12 either alone or as part of a treatment regimen.
* Subjects who were administered any live attenuated vaccines within 30 days prior to first MEDI1191 injection.
* Known allergy or hypersensitivity to any component of MEDI1191 or durvalumab formulations.
* Active or prior documented autoimmune disorders within the past 5 years prior to the first scheduled dose of study treatment except alopecia, hypothyroidism (stable of hormone replacement), chronic skin condition (does not require systemic therapy), and celiac disease (controlled by diet alone).
* Immune-deficiency states - myelodysplastic disorders, marrow failure states, human immunodeficiency virus infection, history of solid organ transplant, bone marrow allograft, or active tuberculosis.
* History of coagulopathy resulting in uncontrolled bleeding or other bleeding disorders.
* Require continuous anticoagulation or antiplatelet therapy (except for ≤ 100 mg acetylsalicylic acid [ASA]) which cannot be interrupted for more than 7 days for IT delivery of MEDI1191.
* Any concurrent chemotherapy, radiotherapy, immunotherapy, biologic or hormonal therapy for cancer.
* Receipt of any conventional or investigational anticancer therapy within 21 days or palliative radiotherapy within 7 days prior to the first dose of study treatment. For subjects who have received prior immunotherapy, the following additional exclusion criteria apply:

  1. Received only one dose of prior immunotherapy agent alone or as part of a combination regimen
  2. Experienced a toxicity that led to permanent discontinuation of prior immunotherapy
  3. All AEs while receiving prior immunotherapy did not resolve to ≤ Grade 1 or baseline prior to screening for this study.
  4. Experienced a ≥ Grade 3 AE (including pneumonitis) or neurologic, ocular, or cardiac AE of any grade while receiving prior immunotherapy.
  5. Required the use of additional immunosuppression other than corticosteroids for the management of an AE, or experienced recurrence of an AE if re-challenged, or is currently requiring a maintenance dose of > 12 mg prednisone or equivalent per day.
* Any toxicity from prior therapy that has not completely resolved to ≤ Grade 1 or baseline at the time of consent.
* Current or prior use of immunosuppressive medication within 14 days prior to the first dose of MEDI1191, except intranasal, topical, inhaled corticosteroids, local steroid injections, systemic corticosteroids at physiologic doses not to exceed 12 mg/day of prednisone or equivalent, or steroids as premedication for hypersensitivity reactions.
* Cardiac exclusions: New York Heart Association Class 3 or 4 congestive heart failure, uncontrolled hypertension, acute coronary syndrome within 6 months.
* Any condition that would interfere with evaluation of the investigational product or interpretation of subject safety or study results.
* Uncontrolled intercurrent illness.
* Untreated, active hepatitis B or C.
* Major surgery within 4 weeks prior to first dose of MEDI1191 or still recovering from prior surgery.
* Subjects with untreated active major depression with suicidal ideation and/or plan.
* Female subjects who are pregnant, lactating, or intend to become pregnant during their participation in this study.

Ages: 18 Years to 101 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2023-08-24 (Actual); Study Completion 2023-08-24 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events (AEs) serious adverse events (SAEs) and dose limiting toxicities (DLTs). | From time of informed consent until 90 days after the last dose of investigational product (MEDI1191 or durvalumab).
  The occurrence of DLTs will be used to establish the maximum tolerated dose (MTD) of MEDI1191.
Objective response rate (ORR) in patients within expansion arms. | Estimated to be from time of informed consent up to 3.5 years.
  The ORR is defined as the proportion of subjects with confirmed response (CR) or confirmed partial response (PR).

SECONDARY OUTCOMES:
Number of advanced solid tumor subjects with adverse events (AEs) serious adverse events (SAEs) and dose limiting toxicities (DLTs). | From time of informed consent until 90 days after the last dose of investigational product (MEDI1191 or durvalumab).
  The occurrence of DLTs will be used to establish the maximum tolerated dose (MTD) of MEDI1191.
Objective response rate (ORR) in advanced solid tumor subjects. | Estimated to be from time of informed consent up to 3.5 years.
  The ORR is defined as the proportion of subjects with confirmed response (CR) or confirmed partial response (PR).
Disease Control Rate (DCR). | Estimated to be from time of informed consent up to 3.5 years.
  The DCR will be estimated by the proportion of disease control. Disease control is defined as CR, PR or stable disease.
Duration of Response (DoR). | Estimated to be from time of informed consent up to 3.5 years.
  The DoR is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first.
Time To Response (TTR). | Estimated to be from time of informed consent up to 3.5 years .
  The TTR is defined as the time from the start of treatment with any investigational product until the first documentation of a subsequently confirmed objective response.
Progression Free Survival (PFS). | Estimated to be from time of informed consent up to 3.5 years.
  PFS will be measured from the start of treatment with any investigational product until the first documentation of disease progression or death due to any cause, whichever occurs first.
Overall Survival (OS). | Estimated to be from time of informed consent up to 3.5 years.
  OS will be measured from the start of treatment with investigational product until death due to any cause.
Maximum observed concentration (Cmax) of MEDI1191 and durvalumab | From first dose of MEDI1191 through to 30 days after last dose of investigational product.
  The endpoints for assessment of PK of MEDI1191 and durvalumab include individual MEDI1191 and durvalumab concentrations in serum at different timepoints after administration.
Area under the concentration-time curve (AUC) of MEDI1191 | From first dose of MEDI1191 through to 30 days after last dose of investigational product.
  The endpoints for assessment of PK of MEDI1191 include MEDI1191 concentrations in serum at different timepoints after administration.
Clearance of MEDI1191 | From first dose of MEDI1191 through to 30 days after last dose of investigational product.
  The endpoints for assessment of PK of MEDI1191 include MEDI1191 concentrations in serum at different timepoints after administration.
Immunogenicity of MEDI1191 | From first dose of MEDI1191 through to 3.5 years after last dose of investigational product.
  The endpoints for assessment of immunogenicity of MEDI1191 include the number and percentage of subjects who develop detectable anti-drug antibodies (ADAs).

CONTACTS AND LOCATIONS:
Overall Officials: MedImmune LCC, Study Director — MedImmune LLC
Locations (9):
- United States (6):
  - Research Site, La Jolla, California
  - Research Site, Los Angeles, California
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Providence, Rhode Island
  - Research Site, Houston, Texas
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Pamplona

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CRS Synopsis Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8510C00001&attachmentIdentifier=d9f71fe2-ef6c-49bd-b277-598cee46b9b1&fileName=CRS_Synopsis_Redacted.pdf&versionIdentifier=
- See also: Study Results — https://www.astrazenecaclinicaltrials.com/study/D8510C00001/